CLINICAL TRIAL: NCT05510804
Title: Ambulante Leitlinienkonforme Intervention im Selbstmanagement für Angststörungen (ALISA)
Brief Title: Efficacy of an App-based CBT Featuring Virtual Reality for Anxiety Disorders
Acronym: ALISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bartosz of Zurowski (Other)
Collaborators: Zentrum für Integrative Psychiatrie (Other)
Responsible Party: Sponsor-Investigator, Bartosz of Zurowski, Principal Investigator, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ 19-187
Record Dates: First submitted 2021-12-07; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Social Phobia; Panic Disorder; Agoraphobia
Keywords: Digital Health Application; Exposure; Virtual Reality; Cognitive Behavior Therapy
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Panic Disorder; Agoraphobia

STUDY DESIGN:
Intervention Model Description: RCT with 2:1 allocation either to Intervention or TAU (low-frequency unstructured contacts with therapist)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALISA (therapist-assisted digital self-help intervention) (Experimental): structured app-based self-help programme with scheduled therapist assistance
  Interventions: Combination Product: ALISA
- TAU (supportive therapist contacts) (Active Comparator): low-frequency supportive therapist contacts
  Interventions: Combination Product: ALISA

INTERVENTIONS:
Combination Product: ALISA — assisted self-help smartphone application featuring virtual reality within a structured CBT programme / low-frequency scheduled therapist assistance
  Other Names: Invirto

SUMMARY:
Primary aim is to evaluate the efficacy of a (minimally) therapist-guided app-based psychotherapy with virtual reality exposure therapy (ALISA) in participants with agoraphobia with or without panic disorder, social anxiety disorder or panic disorder. Participants are diagnosed applying a structured clinical interview by qualified psychologists and then they are randomly allocated to either the intervention group (ALISA) or a control group, receiving supportive psychotherapy while on a waiting list for a structured therapy programme. The investigators hypothesize that participants receiving ALISA compared to controls will present lower levels of anxiety and a higher quality of life at six-month follow-up after start of the intervention, according to Beck Anxiety Inventory (BAI, primary outcome measure) and WHO-QoL, respectively.

DETAILED DESCRIPTION:
Primary aim is to evaluate the efficacy of a (minimally) therapist-guided app-based psychotherapy with virtual reality exposure therapy (ALISA) in participants with agoraphobia (with or without panic disorder), social anxiety disorder or panic disorder. The intervention has been developed by Sympatient GmbH in cooperation with the University of Luebeck, Dept. of Psychiatry. It consists of scheduled therapist assistance, a smartphone-based application consisting of eight CBT-based courses including instructive therapist videos, questionnaires and VR exposure scenarios presented via VR goggles as well as interoceptive exposures.

Participants are diagnosed according to a structured clinical interview (SCID) by experienced and trained clinical psychologists. Then they are randomly allocated to either the intervention group (ALISA) or a control group offered supportive psychotherapy while being on a waiting list for a structured therapy programme of an outpatient unit for patients with anxiety disorders. The investigators hypothesize that participants receiving ALISA - as compared to controls - will present lower levels of anxiety and a higher quality of life at 6-month follow-up after start of the intervention, according to Beck Anxiety Inventory (BAI, primary outcome measure) and WHO-QoL (L-1), respectively. Furthermore, the investigators hypothesize that the reduction of anxiety (ANOVA; group x time) can be shown at 1-year follow up. The investigators expect ALISA to be effective in each of the three disorder-specific therapy schedules (social phobia, panic disorder, agoraphobia w/without panic disorder). Therefore, disorder-specific symptom scales have been additionally adopted: Panic and Agoraphobia Scale (PAS) and Liebowitz Social Phobia Scale. Co-morbid depression and global functioning will be assessed using CGI and GAF as secondary outcome measures, respectively.

The allocation to the groups was conducted on the basis of random numbers generated by Microsoft Excel 2013 and with the restriction that the ratio of intervention to control group participants was 2:1. This unequal randomization was chosen for ethical reasons including a more reliable assessment of adverse events in the intervention group with a higher power. A planned sample size of n = 41 for each of the three diagnoses in the intervention group and n = 21 for each of the three diagnoses in the control group was calculated to detect a significant difference with an effect size of Cohens´s d = 0.9 with a probability of 90% and α = 2.5. Adding an estimated dropout-rate of 20%, each diagnosis group should include n = 49 participants in the intervention group and n = 25 in the control group, resulting in a total of N = 222 participants. (Multiple) imputation will be applied to deal with missing data. Results of Intention to treat analyses and following per protocol analyses will be reported.

Using records of cooperating health insurances, a health economic analysis of the intervention will be performed. Given that patients with untreated anxiety disorders show a markedly increased use of health system, a successful reduction of anxiety, once proven, should have an impact on patient's use of the health system in general (exploratory analysis)

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: Agoraphobia w/without PD (F 40.0, F40.01) OR Panic disorder (F41.0) OR Social anxiety disorder (phobia) (F40.1)
* Smartphone availability

Exclusion Criteria:

* history of stroke or heart attack
* angina pectoris
* cardiac arrhythmia
* untreated high blood pressure
* severe asthma or chronic obstructive pulmonary disease (COPD)
* (supposed) pregnancy
* severe visual impairment
* severe nausea and/or vestibular impairment
* epilepsy
* neuropsychiatric condition (i.e. dementia)
* psychiatric disorder associated with substance abuse
* psychotic disorder
* severe episode of major depression or manic episode
* suicidal ideation or behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) | 6 months after inclusion
  standard self-report instrument (21 items) for anxiety applicable in all three disorders investigated

SECONDARY OUTCOMES:
Change in Clinical Global Impression CGI | through intervention completion, on average month 3
  broadly used measure of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders It is a brief 3-item observer-rated scale for clinical practice and research.
Change in Global Assessment of Functioning (GAF) | through intervention completion, on average month 3
  broadly used and WHO-recommended scale to evaluate an individual's' psychological, social, and occupational functioning (0-100)
Change in WHO QoL L-1 | 6 months after inclusion
  one-item assessment of quality of life
Change in WHO QoL L-1 | 12 months after inclusion
  one-item assessment of quality of life
Change in Beck Anxiety Inventory (BAI) | 12 months after inclusion
  standard self-report instrument (21 items) for anxiety applicable in all three disorders

OTHER OUTCOMES:
Change in Beck Depression Inventory (BDI II) | 6 months after inclusion
  standard self-report instrument (21 items) measuring depressive symptoms
Change in Beck Depression Inventory (BDI II) | 12 months after inclusion
  standard self-report instrument (21 items) measuring depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Zurowski, Principal Investigator — Zentrum für Integrative Psychiatrie, Univ. of Luebeck
Locations (2):
- Germany (2):
  - Zentrum für Integrative Psychiatrie, Univ. of Kiel, Kiel, Schleswig-Holstein
  - Zentrum für Integrative Psychiatrie, Univ. of Lübeck, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No